CLINICAL TRIAL: NCT05714878
Title: Multimodal Prehabilitation for Patients With Resectable Gastric Cancer: A Randomized Controlled Trial
Brief Title: Multimodal Prehabilitation for Resectable Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Kecheng Zhang, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLAGH202212
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Stomach Neoplasm
Keywords: Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Exercise; Nutritional Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation arm (Experimental): Patient receives prehabilitation intervention including exercise, nutrition and psychological support.
  Interventions: Behavioral: aerobic exercise; resistance exercise; nutritional support; psychological support
- Control arm (No Intervention): Patient receives regular care recommended by the WHO without supervision and support.

INTERVENTIONS:
Behavioral: aerobic exercise; resistance exercise; nutritional support; psychological support — Patient with gastric cancer received two weeks of prehabilitation intervention. An individualized exercise program was established according to the FITT (Frequency, Intensity, Time and Type) principle. Aerobic exercise: 3-5 times/week, 30-60 min jogging or brisk walking per time, intensity based on heart rate and modified Borg-scale. Resistance exercise: 2-3 times/week, 10-12 RM per sets, 2-3 sets with 2 min interval rest, seated knee up, knee extension, etc. Nutritional support: 30kcal/kg/d, 1.5mg/kg/d protein, oral nutritional supplement with suggested recipes. Psychological support: provided with guidance on gastric cancer, regular online chat through Wechat, alcohol quitting, smoking cessation and light music.
  Arms: Prehabilitation arm

SUMMARY:
Surgical resection is the mainstay for gastric cancer. Surgical stress response, like insulin resistance and catabolism, is inevitable and is a risk factor for postoperative outcome. To cope with this stress, the enhanced recovery protocol has been proposed and successfully implemented in clinical practice. Recently, prehabilitation have attracted increasingly attention, which is the preoperative part of enhanced recovery pathway. Prehabtilitation are bundles of evidenced elements in order to improve patient's functional capacity. Patients with gastric cancer are usually suffered from nutritional risk, anxiety and frailty. In this trial, we investigate whether multimodal prehabilitation (exercise, nutrition and psychological support) could improve patient's functional status to better tolerate surgical trauma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric cancer, clinical I-III TNM stage (AJCC 8th edition);
* Will receive curative-intent surgery;
* Life expectance > 6 months;

Exclusion Criteria:

* Gastric stump cancer or combined with other malignances;
* NYHA III, NYHA IV;
* Inability to swallow, with gastrostomy, or inability to move because of orthopedic disease or neuromuscular disease;
* Psychiatric disorders, COPD, end-stage hepatic or renal disease, uncontrolled cardiac arhythmia or uncontrolled hypertention;
* Receiving immunosuppressive therapy;
* Emergency surgery because of tumor bleeding or tumor perforation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Duke Activity Status Index before surgery | Duke Activity Status Index score on the day before surgery
  Duke Activity Status Index score is a 12-item self-reported questionnaire that assesses daily activities such as personal care, ambulation, household tasks, and recreation with respective metabolic costs. Duke Activity Status Index score ranges from 0 to 58.2. The higher score indicates the better functional status. Duke Activity Status Index has been recommended by European Society of Cardiology guidelines for functional assessment of patients undergoing non-cardiac surgery.

SECONDARY OUTCOMES:
Morbidity | In postoperative 30 day after gastrectomy
  Postoperative complication
Postoperative hospital stay | During the postoperative 30 day period
  Period from day of surgery to day of discharge from hospital
30-day readmission rate | During the postoperative 30 day period
  Proportion of patients admitted to the hospital after discharge because of complications

CONTACTS AND LOCATIONS:
Overall Officials: Kecheng Zhang, Principal Investigator — Chinese PLA General Hospital First Medical Center
Locations (1):
- Chinese PLA General Hospital First Medical Center, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halvorsen S, Mehilli J, Cassese S, Hall TS, Abdelhamid M, Barbato E, De Hert S, de Laval I, Geisler T, Hinterbuchner L, Ibanez B, Lenarczyk R, Mansmann UR, McGreavy P, Mueller C, Muneretto C, Niessner A, Potpara TS, Ristic A, Sade LE, Schirmer H, Schupke S, Sillesen H, Skulstad H, Torracca L, Tutarel O, Van Der Meer P, Wojakowski W, Zacharowski K; ESC Scientific Document Group. 2022 ESC Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Eur Heart J. 2022 Oct 14;43(39):3826-3924. doi: 10.1093/eurheartj/ehac270. No abstract available. PMID 36017553
- [Background] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252